CLINICAL TRIAL: NCT00396253
Title: A Phase III, Open-Label Study of Tenecteplase for Restoration of Function in Dysfunctional Hemodialysis (HD) Catheters
Brief Title: A Study of Tenecteplase for Restoration of Function in Dysfunctional Hemodialysis (HD) Catheters
Acronym: TROPICS 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N3701g
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Dysfunctional Hemodialysis Catheters
Keywords: HD; TNKase; Hemodialysis; Catheter clearance
MeSH Terms: interventions — Tenecteplase

ARMS (1):
- Tenecteplase (Experimental): At each treatment, subjects had 2 mL (2 mg) of tenecteplase instilled into each lumen of their HD catheter. Subjects could receive up to three treatments with tenecteplase, the first two as part of the initial treatment course and one additional treatment as part of the retreatment (RT) course. The first treatment, followed by a 1-hour dwell time, was given to all subjects at Visit 1. At the end of hemodialysis at Visit 1, eligible subjects had a second treatment instilled for an extended dwell time until the start of Visit 2 (up to 72 hours).
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — 2 mL (2 mg) of reconstituted lyophilized tenecteplase instilled into each lumen of the HD catheter.

SUMMARY:
This was a Phase III, open-label study conducted at 44 centers in the United States, Canada, and Puerto Rico. 223 subjects who required hemodialysis (HD) and had a dysfunctional HD catheter were enrolled in the study.

DETAILED DESCRIPTION:
The study consisted of four visits that corresponded to consecutive HD sessions for each patient, as well as one follow-up visit. Patients could receive up to three treatments with open-label tenecteplase during the study: one or two treatments during an initial treatment course, and eligible patients whose catheter became dysfunctional again within 21 days of the first visit received an additional treatment as part of a retreatment (RT) course.

At Visit 1, patients eligible at the beginning of HD had 2 mL (2 mg) of tenecteplase instilled into each of the two lumens of the HD catheter. After a dwell time of 1 hour, study drug was withdrawn and all subjects underwent HD. The duration of the HD session was not fixed by the study protocol, but rather by the site's HD practice, physician orders, and individual patient response during the session. Patients who did not experience treatment success at the end of Visit 1 had 2 mL (2 mg) of tenecteplase instilled into each lumen of their catheter as part of the initial treatment course. The treatment was left to dwell for an extended time, until the second HD session at Visit 2 (up to 72 hours later). Patients who received extended-dwell tenecteplase had the treatment withdrawn from their catheter at the beginning of Visit 2. Patients underwent HD as prescribed or to the extent possible.

Patients who had treatment success at Visit 1 or Visit 2 and had a recurrence of catheter dysfunction within 21 days of Visit 1 and met the re-treatment eligibility criteria had 2 mL (2 mg) of tenecteplase instilled into each lumen, followed by a 1-hour dwell time at re-treatment Visit 1.

ELIGIBILITY:
Inclusion Criteria: for the Study

* Clinically stable, in the opinion of the investigator
* Use of a cuffed, tunneled HD catheter
* HD prescribed at a blood flow rate (BFR) of ≥300 mL/min
* Baseline BFR (at any time during the first 60 minutes of HD) of <300 mL/min at an associated pre-pump negative arterial pressure in the range between and including -240 mmHg and -280 mmHg
* Baseline BFR (at any time during the first 60 minutes of HD) at least 25 mL/min below the prescribed BFR
* Demonstrated BFR of ≥300 mL/min (using catheter lines in the customary direction) at an arterial pressure in the range of 0 to -280 mmHg in at least one HD session in the 14 days prior to Visit 1
* Anticipated use of the same catheter for at least four consecutive HD sessions, on the same type and model of HD apparatus
* Able to have fluids infused at the volume necessary to instill study drug into the HD catheter

Exclusion Criteria: for the Study

* HD catheter with sustainable BFR of ≥300 mL/min following subject repositioning
* HD catheter inserted <2 days prior to screening
* Evidence of a mechanical, non-thrombotic cause of HD catheter dysfunction (e.g., kink in the catheter or suture constricting the catheter) or dysfunction caused by known fibrin sheath
* Use of an implantable port
* HD catheter that is internally coated with any therapeutic agent (e.g., the Decathlon™ Gold catheter)
* Anticipated use of catheter for any other type of diagnostic or therapeutic procedure (i.e., other than HD) during study drug treatment
* Previously treated in this study or any tenecteplase catheter clearance trial
* Use of any investigational drug or therapy (defined as any drug or therapy that is not FDA approved) within 28 days prior to screening
* Use of a fibrinolytic agent (e.g. alteplase, tenecteplase, reteplase, or urokinase) within 7 days prior to Visit 1
* Known to be pregnant or breastfeeding at screening or at Visit 1
* Known bacteremia or known or suspected infection in the HD catheter
* Known history of any of the following: intracranial hemorrhage (within the previous 3 years), intracranial aneurysm, or arteriovenous malformation
* Use of heparin (unfractionated or low molecular weight) or other anticoagulants (e.g., for the treatment of heparin-induced thrombocytopenia) within 24 hours prior to Visit 1, except for heparin used only during HD or for prophylaxis (e.g., heparin lock or deep vein thrombosis prophylaxis)
* Subjects treated with warfarin only: international normalized ratio (INR) >3.0 within 7 days prior to Visit 1, or a target INR range that allows for an INR >3.0
* Initiation of or increase in dose of Plavix® (clopidogrel bisulfate) within 7 days prior to Visit 1
* Hemoglobin ≥12.0 g/dL if on an erythropoiesis-stimulating agent (e.g., darbepoetin or erythropoietin) and the dose of the erythropoiesis-stimulating agent has not been held or reduced per institutional policy
* At high risk for bleeding events or embolic complications (i.e., recent pulmonary embolus, deep vein thrombosis, endarterectomy, or clinically significant right-to-left shunt) in the opinion of the investigator, or with known condition for which bleeding constitutes a significant hazard
* BFR of <300 mL/min because of symptomatic hypotension
* Uncontrolled hypertension in the opinion of the investigator
* Known hypersensitivity to tenecteplase or any component of the formulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gillespie, MD, FASN, Study Director — Quintiles, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenecteplase: At each treatment, patients had 2 mL (2 mg) of tenecteplase instilled into each lumen of their HD catheter. Patients could receive up to three treatments with tenecteplase, the first two as part of the initial treatment course and one additional treatment as part of the retreatment (RT) course. The first treatment, followed by a 1-hour dwell time, was given to all patients at Visit 1. At the end of hemodialysis at Visit 1, eligible patients had a second treatment instilled for an extended dwell time until the start of Visit 2 (up to 72 hours).
Period: Overall Study
Arm/Group | Tenecteplase
Started | 223
Completed | 210
Not Completed | 13
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 7
Not completed — Death | 3
Not completed — Physician Decision | 1
Not completed — Change in eligibility status | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tenecteplase
Number analyzed (Participants) | 223
Age, Customized [Number; unit: participants]
  < 17 years | 1
  >= 17 years to < 65 years | 120
  >= 65 years | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (16.3)
Gender [Count of Participants; unit: Participants]
  Female | 124
  Male | 99

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Treatment Success With Respect to Blood Flow Rate (BFR) at Visit 1
Description: Treatment success is defined as Blood Flow Rate (BFR) ≥ 300 mL/min and an increase of ≥ 25 mL/min from baseline BFR (without reversal of lines), at an associated arterial pressure in the range of 0 to -280 mmHg, 30 (± 10) minutes prior to the end of hemodialysis and at the end of hemodialysis.
Time Frame: Visit 1 (the first hemodialysis session in which treatment was administered). BFR was measured at the beginning of hemodialysis (Baseline measurement) and at 30 minutes prior to the end of hemodialysis and at the end of hemodialysis.
Population: Modified intent to treat (MITT) population, consisting of all enrolled patients who received at least one dose of study drug (tenecteplase).
Measure: Number; unit: Percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 223
Percentage of participants | 34.1

2. Primary Outcome: Targeted Adverse Events From the Initial Study Drug Administration Through the Start of Visit 2 or Until Instillation of Extended-Dwell Tenecteplase
Description: The primary outcome measure was the number of targeted adverse events, occurring from initial study drug administration through the end of Visit 1 (prior to administration of open-label, extended-dwell tenecteplase) or, for subjects who did not receive open-label, extended-dwell tenecteplase, from initial study administration through the start of Visit 2. Targeted adverse events were defined as intracranial hemorrhage, major bleeding and embolic events, thrombosis, Catheter-related blood stream infection (CRBSIs), and catheter-related complications.
Time Frame: From initial study drug administration to the end of Visit 1 (prior to administration of open-label, extended-dwell tenecteplase) or, for patients who did not receive extended-dwell tenecteplase, from initial study administration to the start of Visit 2.
Population: Modified intent to treat (MITT) population
Measure: Number; unit: Events
Arm/Group | Tenecteplase
Number analyzed (Participants) | 223
Events
  Intracranial hemorrhage | 0
  Major bleeding | 0
  Embolic event | 0
  Thrombosis | 1
  Catheter-related blood stream infection | 2
  Catheter-related complication | 0

3. Secondary Outcome: Percentage of Participants Who Maintained Catheter Function at Visits 2 and 3
Description: For patients with treatment success at Visit 1 or Visit 2, maintenance of catheter function at subsequent visits was defined as a BFR ≥ 300 mL/min and an increase of ≥ 25 mL/min from baseline BFR (without reversal of lines), at an associated target arterial pressure in the range of 0 to -280 mmHg at the beginning of that HD session (within the first 30 minutes).
Time Frame: Maintenance BFR measurements were taken at the beginning of HD at Visit 2 (2nd consecutive HD session, within 72 hours of Visit 1) and Visit 3 (3rd consecutive HD session, within 72 hours of Visit 2).
Population: Modified intent to treat (MITT) population, who had treatment success at Visit 1. The n equals the number of subjects who had treatment success at Visit 1 and had assessment of catheter function for the given visit or who had a missing assessment due to starting the Retreatment course.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 76
percentage of participants
  Visit 2 (n=72) | 69.4 [58.8 to 80.1]
  Visit 3 (n=71) | 62.0 [50.7 to 73.3]

4. Secondary Outcome: Percentage of Participants With Urea Reduction Ratio ≥ 65% at Visit 1
Description: The urea reduction ratio (URR) was calculated from measurements of blood urea nitrogen (BUN) as follows:
  (Pre-treatment BUN) - (Post-HD BUN) * 100% / (Pre-treatment BUN)
  Pre-treatment URR was assessed within 30-60 minutes after the initiation of HD and does not represent a true baseline value.
Time Frame: At Visit 1 (first hemodialysis session in which treatment was administered) samples for blood urea nitrogen measurements were taken at the beginning of HD (prior to treatment administration) and after HD was completed.
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 223
percentage of participants | 23.8 [18.2 to 29.4]

5. Secondary Outcome: Percentage of Participants With Urea Reduction Ratio ≥ 65% at Visit 2
Description: The urea reduction ratio (URR) at Visit 2 was calculated for those participants who did not receive extended-dwell tenecteplase at Visit 1 from measurements of blood urea nitrogen (BUN) as follows:
  (Pre-HD BUN) - (Post-HD BUN) * 100% / (Pre-HD BUN)
Time Frame: At Visit 2 (2nd consecutive HD session, within 72 hours of Visit 1) samples for blood urea nitrogen measurements were taken prior to HD and after HD was completed.
Population: Modified intent to treat (MITT) population who did not receive extended-dwell tenecteplase at Visit 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 107
percentage of participants | 34.6 [25.6 to 43.6]

6. Secondary Outcome: Change in Blood Flow Rate From Baseline to the End of Hemodialysis at Visit 1
Description: Change in Blood flow rate (BFR) is the BFR at the end of HD for Visit 1 - BFR at Baseline.
Time Frame: Baseline (beginning of HD at Visit 1) to the end of HD at Visit 1.
Population: Modified intent to treat (MITT) population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Tenecteplase
Number analyzed (Participants) | 223
mL/min | 81.9 (123.84)

7. Secondary Outcome: Percentage of Participants Who Failed Treatment at Visit 1 With Treatment Success at Visit 2
Description: Patients who failed treatment at Visit 1 and were treated with extended-dwell tenecteplase were analyzed for Treatment Success at Visit 2. Treatment success at Visit 2 was defined as a BFR ≥ 300 mL/min, without line reversal, and increase of ≥ 25 mL/min from baseline BFR, at an associated target arterial pressure in the range of 0 to -280 mmHg, 30 (± 10) minutes prior to the end of HD and at the end of HD.
Time Frame: BFR was measured 30 minutes before the end of HD and at the end of HD at Visit 2 (2nd consecutive HD session, within 72 hours of Visit 1). Baseline BFR was measured at the beginning of HD at Visit 1.
Population: Subjects in the MITT Population who were Treated with Extended-Dwell Tenecteplase at Visit 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 116
percentage of participants | 49.1 [40.0 to 58.2]

8. Secondary Outcome: Percentage of Participants Who Failed Treatment at Visit 1 With a Urea Reduction Ratio ≥ 65% at Visits 2 and 3
Description: Patients who experienced treatment failure at the end of Visit 1 and were eligible for and treated with extended-dwell tenecteplase at Visit 1 were assessed for Urea Reduction Ratio (URR) at Visits 2 and 3. URR was calculated from blood urea nitrogen (BUN) measurements according to the following:
  (Pre-HD BUN) - (Post-HD BUN) * 100% / (Pre-HD BUN)
Time Frame: Blood urea nitrogen measurements were taken prior to HD and at the end of HD at Visits 2 (2nd HD session, within 72 hours after visit 1) and 3 (3rd HD session, within 72 hours of Visit 2)
Population: Subjects in the MITT Population who were Treated with Extended-Dwell Tenecteplase at Visit 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tenecteplase
Number analyzed (Participants) | 116
percentage of participants
  URR ≥ 65% at Visit 2 | 42.2 [33.3 to 51.2]
  URR ≥ 65% at Visit 3 | 33.6 [25.0 to 42.2]

9. Secondary Outcome: Change in Blood Flow Rate From Baseline to the End of HD at Visit 2
Description: Change in Blood flow rate (BFR) is the BFR at the end of HD for Visit 2 - BFR at Baseline.
Time Frame: Baseline (beginning of HD at Visit 1) to the end of HD at Visit 2 (2nd consecutive HD session, within 72 hours of Visit 1).
Population: Subjects in the MITT Population Treated with Extended-Dwell Tenecteplase at Visit 1
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Tenecteplase
Number analyzed (Participants) | 116
mL/minute | 117.1 (139.96)

ADVERSE EVENTS:
Time Frame: Begins at initiation of study treatment and ends upon completion of the second visit following the last administration of study treatment or at early termination from the study, whichever is earlier.
Description: MITT population.
  Note: The incidence of each AE/SAE is reported as the number of participants experiencing the event, not the number of occurrences for each AE/SAE.
Arm/Group | Tenecteplase
Serious Adverse Events (participants affected / at risk) | 9/223
Other Adverse Events (participants affected / at risk) | 36/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=223)
Anaemia (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Catheter Bacteraemia (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Infected Skin Ulcer (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=223)
Nausea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Catheter Site Erythema (General disorders) | 1
Catheter Site Pain (General disorders) | 1
Chest Pain (General disorders) | 1
Chills (General disorders) | 1
Feeling Hot (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Abdominal Abscess (Infections and infestations) | 1
Central Line Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Device Breakage (Injury, poisoning and procedural complications) | 1
Body Temperature Increased (Investigations) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3
Haemodynamic Instability (Vascular disorders) | 2
Hot Flush (Vascular disorders) | 1
Venous Thrombosis Limb (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.